CLINICAL TRIAL: NCT02995252
Title: An Omnibus Protocol to Characterize Patients With Hepatitis B and C (the HOPE Study) With Hepatitis B Treatment Sub-study
Brief Title: The HOPE Study: Characterizing Patients With Hepatitis B and C
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Lydia Tang, MD, University of Maryland, Baltimore
Other Study IDs: HP-00063191
Record Dates: First submitted 2016-12-13; First posted 2016-12-16 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hepatitis B， Chronic; Hepatitis C
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis C | interventions — Blood Specimen Collection; tenofovir alafenamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — one sample of blood is collected and stored for future analysis of genetic markers relevant to disease outcomes.
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Hepatitis C infection: Participants with chronic hepatitis C infection; includes both hepatitis C mono infected and hepatitis C-HIV coinfected. Participants will attend study visits for research blood draws (once a year with optional additional visits), and a one-time optional knowledge questionnaire. No drugs will be given to this group.
  Interventions: Other: Blood draws; Other: Knowledge Index Questionnaire
- Group 2: Hepatitis B infection: Participants with chronic hepatitis B: includes patients with hepatitis B with and without hepatitis C and/or HIV. Participants will attend study visits for research blood draws (once a year with optional additional visits), and a one-time optional knowledge questionnaire. Participants who are already taking hepatitis B treatment are eligible.
  Hepatitis B treatment sub-study: In this treatment sub-study, participants with hepatitis B monoinfection will receive tenofovir alafenamide (TAF) pill once a day for 2 years with study visits every 3 months. Liver transient elastography will be reviewed or obtained. In addition, approximately 40 participants will be invited to undergo optional liver biopsies at the start, end of year 1 and end of year 2 of the sub-study.
  Interventions: Other: Blood draws; Drug: Tenofovir Alafenamide; Other: Knowledge Index Questionnaire; Other: Liver transient elastography (FibroScan); Procedure: Liver Biopsy

INTERVENTIONS:
Other: Blood draws
Drug: Tenofovir Alafenamide — 25 mg tablet, once a day by mouth.
  Groups: Group 2: Hepatitis B infection
Other: Knowledge Index Questionnaire
Other: Liver transient elastography (FibroScan) — Participants of the hepatitis B treatment sub-study may have FibroScans completed at baseline, during the study with liver enzyme normalization, and at the end of the study.
  Groups: Group 2: Hepatitis B infection
Procedure: Liver Biopsy — 40 participants of the hepatitis B treatment sub-study will have liver biopsies prior to starting tenofovir alafenamide, and at years 1 and 2 of receiving treatment.
  Groups: Group 2: Hepatitis B infection

SUMMARY:
This is an observational, longitudinal, prospective study for sample collection and evaluation for future therapy or disease progression of chronic hepatitis B and C. Participants will be seen on an annual basis with optional additional visits for up to 10 years and provide samples for research and evaluation of disease progression. In addition, there is a longitudinal sub-study for treatment of hepatitis B that will involve 2 years of treatment with tenofovir alafenamide and blood collections with optional liver biopsies.

DETAILED DESCRIPTION:
Hepatitis B virus chronically infects 350 million people worldwide and over one million Americans and approximately 4.1 million individuals (1.6%) in the US population have been infected with hepatitis C. These infections are the leading cause of end-stage liver disease, cancer and indication for liver transplantation in the world. Both can be transmitted sexually, perinatally and percutaneously. Coinfected with human immunodeficiency virus (HIV) accelerates the progression of liver disease, and due to shared modes of transmission, chronic hepatitis B and C disproportionately affect people living with HIV.

The primary objective of this study is to Identify people with viral hepatitis and providing linkage to care and future therapy with evaluation of disease progression; as well as characterizing those with hepatitis B and those treated for hepatitis C with directly acting antivirals over the course of 10 years.

The study, including a participant questionnaire and phlebotomy, will be administered on-site at clinical facilities in the District of Columbia and Maryland, and at the Institute of Human Virology at the University of Maryland, Baltimore. The cohort will be designed to study research questions with respect to liver disease, disease pathogenesis using genomics, proteomics, and immunologic disease models. Secondary objectives include study of the immunopathogenesis of hepatitis B and C disease progression. In addition, this is an invaluable opportunity to evaluate the long term effects of hepatitis C clearance with direct acting antivirals, along with biomarker profile(s) for diagnosis and outcome. Moreover, this will serve as a catchment protocol to select appropriate participants for novel hepatitis B and C therapeutic trials.

This study includes a standard-of-care treatment sub-study for patients with hepatitis B. In this sub-study, participants will receive an approved nucleos(t)ide analogue prospectively observed on therapy for change in liver fibrosis.

The integrated clinics will provide an optimal environment for the adherence and engagement of medical care and education in decreasing transmission risks of infection. The study will establish a blood and specimen repository for participants and include a research database that will be used prospectively to test future hypotheses.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Hepatitis B and/or C-infected; or history of hepatitis B infection, but cleared; or hepatitis C infection and successfully treated with direct acting antiviral agents, with or without HIV infection; or healthy volunteer without history of HBV and/or C, nor HIV
3. Willing to have samples stored for future research
4. Must have an identifiable primary care provider or be in the process of establishing a primary care provider
5. Willing to undergo HIV testing if not recently documented
6. Inclusion in the HBV treatment sub-study will be dependent on eligibility to receive nucleos(t)ide analogue therapy according to standard-of-care.

Exclusion Criteria:

1. Unable to comply with research study visits
2. Poor venous access not allowing screening laboratory collection
3. Have any condition that the investigator considers a contraindication to study participation.
4. HBV monoinfected participants with any contraindications to HBV treatment with nucleos(t)ide analogues will be ineligible to participate in the HBV treatment sub-study.
5. Pregnant or breastfeeding women will not be eligible to participate in the HBV treatment sub-study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with chronic hepatitis B and/or C, with or without HIV infection. Or people who have cleared hepatitis B infection, or been treated for hepatitis C infection with direct acting antiviral agents.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2014-12; Primary Completion 2034-07 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Change in liver stiffness among participants with chronic hepatitis B infection | 2 years
  Participants will be provided with the nucleotide analogue, tenofovir alafenamide. Change in liver stiffness as measured by transient elastography (FibroScan) before starting tenofovir alafenamide, at time of liver enzyme normalization, and at 2 years of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Tang, MBChB, Principal Investigator — Institute of Human Virology, University of Maryland School of Medicine
Locations (2):
- United States (2):
  - Institute of Human Virology, University of Maryland School of Medicine, Baltimore, Maryland
  - Dr Huong Dang, Medical Practice, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No